CLINICAL TRIAL: NCT00635557
Title: Dose Finding Phase 1 Study of the Treatment of Recurrent/Relapsed Glioblastoma Multiforme With MPC-6827 in Combination With Carboplatin
Brief Title: Phase 1 Study of MPC-6827 and Carboplatin in Recurrent/Relapsed Glioblastoma Multiforme
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Myrexis Inc. (Industry)
Responsible Party: Andrew P. Beelen, MD / Sr. Director of Clinical Research, Myrexis Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPC-6827-07-004; MPC-6827 GBM
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Last update posted 2011-03-25 (Estimated); Status verified 2011-03

CONDITIONS: Glioblastoma Multiforme
Keywords: Recurrent; Relapsed; Glioblastoma; Multiforme
MeSH Terms: conditions — Glioblastoma; Recurrence | interventions — verubulin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: MPC-6827 + Carboplatin — MPC-6827 at 2.1mg/m2, 2.7mg/m2 or 3.3mg/m2 administered by intravenous infusion over 2 hours once weekly for three weeks in a 4 week cycle. Carboplatin at AUC4 administered by intravenous infusion over 1 hour on Day 1 of each 4 week cycle.

SUMMARY:
This is an open-label, dose finding, multiple-dose study in subjects with recurring/relapsing glioblastoma multiforme. Three dose levels of MPC-6827 will be administered with carboplatin to three separate cohorts. Study endpoints will include determination of the maximum tolerated dose, dose limiting toxicities, and evaluation of evidence of anti-tumor activity of MPC-6827 when given with carboplatin.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven WHO Grade IV glioblastoma multiforme at time of diagnosis or relapse
* Prior treatment with radiotherapy and temozolomide
* Evidence of measurable recurrent or residual primary tumor by contrast-enhanced MRI
* Be a minimum of 4 weeks since prior surgical resection, major surgical procedure, radiation therapy or cytotoxic chemotherapy (6 weeks since prior BCNU or CCNU)
* Have a Performance Scale of Karnofsky > 60%, ECOG < 2 or WHO < 2
* If steroids are needed, be on a stable or decreasing dose of steroids for at least 1 week

Exclusion Criteria:

* Hypersensitivity to Cremophor EL
* Have evidence of current/active intratumor hemorrhage by MRI
* Have greater than second relapse
* Have had prior treatment with platinum-based chemotherapy
* Have cardiovascular disease
* Have cerebrovascular disease
* Have uncontrolled hypertension
* Have a cardiac ejection fraction < 50%
* Have Troponin-I elevated above the normal range

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-10 (Actual); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | After each cohort is enrolled and all subjects have completed 1 cycle

SECONDARY OUTCOMES:
Pharmacokinetics | Cycle 1 only
Antitumor activity | Screening, end of each cycle, end of study

CONTACTS AND LOCATIONS:
Overall Officials: Andrew P. Beelen, MD, Study Director — Myrexis Inc.
Locations (5):
- United States (5):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - Mt. Sinai School of Medicine, New York, New York
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah